CLINICAL TRIAL: NCT05982366
Title: distAl vs. coNventional Transradial Access for coRonary procEdures Study (ANTARES)
Brief Title: Feasibility and Safety of the Routine Distal Transradial Approach
Acronym: ANTARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Łukasz Koziński (Other)
Responsible Party: Sponsor-Investigator, Łukasz Koziński, Principal Investigator Łukasz Koziński, Indywidualna Praktyka Lekarska Lekarz Łukasz Koziński, Indywidualna Praktyka Lekarska Lekarz Łukasz Koziński
Organization: Indywidualna Praktyka Lekarska Lekarz Łukasz Koziński (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AntaresStudy01
Record Dates: First submitted 2023-06-21; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Vascular Access Complication; Radial Artery; Coronary Artery Disease; Puncture; Coronary Angiography
Keywords: radial artery; distal transradial approach; access complication; anatomical snuffbox
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal transradial approach (Experimental): Distal transradial approach as the default strategy
  Interventions: Other: distal radial artery acess side
- Conventional transradial approach (Active Comparator): Conventional transradial approach as the default strategy
  Interventions: Other: conventional radial artery acess side

INTERVENTIONS:
Other: distal radial artery acess side — coronary procedure (coronary angiography and/or coronary angioplasty) by the distal radial artery in the anatomical snuffbox area
  Other Names: dTRA
  Arms: Distal transradial approach
Other: conventional radial artery acess side — coronary procedure (coronary angiography and/or coronary angioplasty) by the forearm radial artery in the anatomical snuffbox area
  Other Names: cTRA
  Arms: Conventional transradial approach

SUMMARY:
The distal transradial approach (dTRA) via the anatomical snuffbox is hypothesized to be more beneficial than the conventional transradial access (cTRA) in patients undergoing coronary procedures. This prospective single-center randomized trial was designed to investigate the safety, efficacy, and various ultrasound parameters of dTRA.

DETAILED DESCRIPTION:
Transradial approach (TRA) has emerged in most countries as a default strategy in urgent and elective coronary procedures. The advantages of TRA compared to the transfemoral access encompass a reduction of mortality, complications, and cost as well as improvement of patient's comfort. The aim of the present study (ANTARES, distAl vs coNventional Transradial Access for coRonary procEdures Study) was to assess the feasibility, safety and various ultrasound parameters of dTRA in the anatomical snuffbox as the first-line strategy, in comparison with cTRA, in patients undergoing coronary angiography (CAG) and percutaneous coronary intervention (PCI). The study is a non-inferiority, randomized controlled trial. There are two arms: distal transradial access and conventional transradial approach.

400 patients were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for CAG and/or PCI

Exclusion Criteria:

* ST-elevation myocardial infarction
* sudden cardiac arrest
* hemody-namic instability
* chronic kidney disease (stages 4-5)
* forearm artery occlusion
* previous unsuccessful ipsilateral TRA
* unfavorable RA diameter
* ultrasound unavailability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The primary composite endpoint consisted of rate of access crossover, rate of major adverse cardiovascular events (MACE) and rate of access-related vascular complications. | up to 24 hours
  Access crossover from unsuccessful random arterial access (if the initial access point fails) to another one.
  Access-related complications after the procedure measured with Doppler Ultrasound (included radial artery occlusion, significant hematoma (EASY classification grade III-V), arteriovenous fistula, pseudoaneurysm, perforation and spasm).
  MACE definied as myocardial infarction, stroke, urgent revascularization, all-cause death.

SECONDARY OUTCOMES:
efficacy endpoint: rate of access crossover | during the procedure index
  Access crossover from unsuccessful random arterial access (if the initial access point fails) to another one.
safety endpoint: patients' discomfort evaluated during access performance | during the procedure
  physical discomfort at the time of vascular access performance was assessed using a numerical scale (0/1/2/3 - respectively no/mild/moderate/severe discomfort)
efficacy endpoint: duration of access performance | during the procedure index
  (measured from the time of skin puncture with local anesthetic to the successful sheath insertion confirmed by an outflow of arterial blood)
safety endpoint: access-site vascular complications | after 24 hours post procedure
  it is composed by the rate of radial artery occlusion, significant hematoma (EASY classification grade III-V), arteriovenous fistula, pseudoaneurysm, perforation and spasm; measured with Doppler Ultrasound

OTHER OUTCOMES:
Access-time | during procedure
  counted from local anesthesia to successful insertion of the sheath
radial artery size | before the procedure, 24 hours and 60 days after the procedure
  parameter measured by Doppler Ultrasound at the access point
radial artery velocity | before the procedure, 24 hours and 60 days after the procedure
  parameter measured by Doppler Ultrasound at the access point

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Koziński, MD, Study Chair — Indywidualna Praltyka Lekarska Lekarz Łukasz Koziński
Locations (1):
- Szpital Specjalistyczny, Chojnice, Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: No